CLINICAL TRIAL: NCT00958646
Title: Identification of Biomarkers for Investigating Osteopathic Manipulative Treatment
Brief Title: Biomarkers of the Response to Osteopathic Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Kristie Grove Bridges, West Virginia School of Osteopathic Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KB081209; 09-12-580
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: OMT; biomarker; Manipulation, osteopathic
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic Manipulation (Experimental): Standardized OMT procedure
  Interventions: Other: Osteopathic Manipulation
- Placebo (Placebo Comparator): Light touch placebo procedure
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Osteopathic Manipulation — Standardized rib raising protocol
  Arms: Osteopathic Manipulation
Other: Placebo — Light touch control procedure
  Arms: Placebo

SUMMARY:
The purpose of this study is to identify non-invasive biomarkers of the physiologic response to Osteopathic Manipulative Treatment (OMT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 21 and 60

Exclusion Criteria:

* Eating or drinking anything but water or chewing gum within an hour of the appointment
* Rib fracture
* History of unstable cardiac arrhythmia or symptoms related to the chest cavity (difficulty breathing, chest pain)
* Symptoms suggestive of bowel obstruction (abdominal bloating with pain, nausea and vomiting, diarrhea)
* Pregnancy
* History of Sjogren's Syndrome

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Salivary amylase levels | baseline, 10 minutes post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kristie G Bridges, PhD, Principal Investigator — West Virginia School of Osteopathic Medicine
Locations (1):
- West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia, United States